CLINICAL TRIAL: NCT00749398
Title: Atlas of the Evolution of Psoriasis Lesions Under Remicade® : A Dynamic Standardized Photographic Library of Moderate to Severe Psoriasis Subjects Treated With Infliximab
Brief Title: Photographic Library of Moderate to Severe Psoriasis Subjects Treated With Infliximab (Study P05047)
Acronym: PHODYPSO
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P05047
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infliximab: Subjects with moderate-to-severe psoriasis who are treated with infliximab in daily clinics according to local country regulations and reimbursements.
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — According to local country regulations.
  Other Names: Remicade; SCH 215596

SUMMARY:
This is a national, multi-center, observational, prospective photographic atlas study in subjects who are treated with infliximab for moderate-to-severe psoriasis in daily clinic according to local country regulations and reimbursement.

DETAILED DESCRIPTION:
Subjects will enter this study using a non-probability sampling method.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age >=18 with moderate-to-severe psoriasis.
* Patient for whom the physician has decided to initiate psoriasis treatment with infliximab in accordance with the terms of the European labeling.
* Patient must demonstrate his/her willingness to participate in the observational study by signing a written consent.

Exclusion Criteria:

* Patient unable to understand and answer a self administered questionnaire.
* No specific non-inclusion criteria will be applied to eligible patients.
* Contradiction and/or Precaution listed in the Summary of Product Characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation to the observational study will be proposed to Dermatology departments by the medical department of the sponsor. Subjects with moderate-to-severe psoriasis initiating infliximab in accordance with the terms of the European label will be asked to participate.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: Participants with moderate-to-severe psoriasis initiating infliximab in accordance with the terms of the European label were asked to participate in this observational study.
Period: Overall Study
Arm/Group | Infliximab
Started | 124 (Nine participants were excluded because they did not fulfill the inclusion criteria.)
Completed | 71
Not Completed | 53
Not completed — Lack of Efficacy | 7
Not completed — Adverse Event | 4
Not completed — Serious adverse event | 11
Not completed — Withdrawal by Subject | 17
Not completed — Lost to Follow-up | 11
Not completed — Reason not specified | 2
Not completed — Unknown reason | 1

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Static Photographic Physician Global Assessment (PGA) Score as Assessed by Two Dermatologists
Description: Digital pictures of each participant's whole body were taken at each visit. Static PGA was assessed by two dermatologists on the basis of these pictures at a single point in time. The mean of the two readings from the dermatologists was used. Static PGA score ranged from 0 (no psoriasis) to 5 (extreme psoriasis). The higher the number, the more severe the psoriasis was.
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Visit 1 (n=117) | 3.15 (1.02)
  Visit 2 (n=102) | 2.77 (0.98)
  Visit 3 (n=96) | 2.08 (1.01)
  Visit 4 (n=86) | 1.76 (0.95)
  Visit 5 (n=69) | 1.49 (0.86)
  Visit 6 (n=67) | 1.72 (1.04)

2. Secondary Outcome: Static PGA Score as Assessed by the Investigator
Description: Static PGA was assessed at each visit by the investigator. Static PGA score ranged from 0 (no psoriasis) to 5 (extreme psoriasis). The higher the number, the more severe the psoriasis was.
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Visit 1 (n=124) | 3.84 (0.80)
  Visit 2 (n=111) | 3.21 (0.90)
  Visit 3 (n=101) | 2.27 (1.11)
  Visit 4 (n=91) | 1.92 (1.17)
  Visit 5 (n=81) | 1.72 (1.21)
  Visit 6 (n=74) | 2.03 (1.33)

3. Primary Outcome: Dynamic Photographic PGA Score as Assessed by Two Dermatologists
Description: The dynamic PGA score resulted from the comparison of two sets of pictures/visits. The dynamic PGA was scored twice, at the middle and at the end of the observation period (comparison between picture sets of Week 0 (Visit 1) and Week 14 (Visit 4) visits and comparison between picture sets of Week 0 (Visit 1) and Week 30 (Visit 6) visits. Dynamic PGA was assessed by two dermatologists and the mean of the two readings was used. Clinical improvement was measured with a 10 centimeter (cm)-visual analogue scale (VAS) ranging from 0 (no improvement) to 10 (disappearance of lesions).
Time Frame: Week 0 (Visit 1), Week 14 (Visit 4), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Change between Visit 1 and Visit 4 (n=80) | 7.05 (2.32)
  Change between Visit 1 and Visit 6 (n=54) | 7.7 (2.09)

4. Secondary Outcome: Dynamic PGA Score as Assessed by the Investigator
Description: The dynamic PGA was scored twice, at the middle and at the end of the observation period. Clinical improvement from Baseline (Visit 1) was evaluated with a 10 cm-VAS ranging from 0 (no improvement) to 10 (disappearance of lesions) at the Week 14 (Visit 4) and Week 30 (Visit 6) visits.
Time Frame: Week 0 (Visit 1), Week 14 (Visit 4), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Change between Visit 1 and Visit 4 (n=88) | 7.27 (2.63)
  Change between Visit 1 and Visit 6 (n=70) | 7.28 (3.04)

5. Secondary Outcome: Percent Body Surface Area (BSA) Involved With Psoriasis
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5),Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Percent BSA Involved with Psoriasis
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Percent BSA Involved with Psoriasis
  Visit 1 (n=123) | 42.33 (27.12)
  Visit 2 (n=111) | 34.86 (25.95)
  Visit 3 (n=99) | 22.95 (23.84)
  Visit 4 (n=91) | 16.86 (21.42)
  Visit 5 (n=80) | 10.84 (14.17)
  Visit 6 (n=74) | 14.12 (19.26)

6. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score
Description: PASI ranged from 0 (no symptoms) to 72 (very marked symptoms) and assessed 3 clinical signs within each area (head, arms, trunk, and legs): erythema (redness), induration (thickness), and desquamation (scaling).
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Visit 1 (n=124) | 21.92 (15.02)
  Visit 2 (n=109) | 12.95 (10.23)
  Visit 3 (n=101) | 8.00 (8.83)
  Visit 4 (n=90) | 6.38 (7.60)
  Visit 5 (n=81) | 5.33 (6.41)
  Visit 6 (n=74) | 7.17 (8.92)

7. Secondary Outcome: Nail Psoriasis Severity Index (NAPSI) Score
Description: The nail was divided with imaginary horizontal and longitudinal lines into quadrants. Each nail was given a score for nail bed psoriasis (0-4) and nail matrix psoriasis (0-4) depending on the presence of any of the features of nail psoriasis in that quadrant. Each nail was evaluated, and the sum of all the nails was the total NAPSI score. The sum of the scores from all nails ranged from 0 (no psoriasis) to 80 (psoriasis present in all 4 quadrants of all 10 nails).
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Visit 1 (n=86) | 28.74 (23.19)
  Visit 2 (n=75) | 27.08 (23.35)
  Visit 3 (n=70) | 22.17 (21.95)
  Visit 4 (n=64) | 18.64 (19.95)
  Visit 5 (n=53) | 17.53 (20.83)
  Visit 6 (n=52) | 15.67 (17.59)

8. Secondary Outcome: Static PGA Score as Assessed by the Participant
Description: Participants assessed their psoriasis at Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), and Week 30 (Visit 6) according to the Static PGA score, which ranged from 0 (no psoriasis) to 5 (extreme psoriasis). The higher the number, the more severe the psoriasis was.
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Visit 1 (n=121) | 4.02 (0.9)
  Visit 2 (n=101) | 3.35 (0.98)
  Visit 3 (n=96) | 2.5 (1.25)
  Visit 4 (n=87) | 2.24 (1.27)
  Visit 5 (n=77) | 1.9 (1.27)
  Visit 6 (n=71) | 2.2 (1.48)

9. Secondary Outcome: Dynamic PGA Score as Assessed by the Participant
Description: as for outcome 4
Time Frame: Week 0 (Visit 1), Week 14 (Visit 4), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Change between Visit 1 and Visit 4 (n=80) | 6.91 (2.57)
  Change between Visit 1 and Visit 6 (n=70) | 6.56 (3.32)

10. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score
Description: DLQI ranged from 0 (no effect on participant's life) to 30 (extremely large effect on participant's life) and was computed by summing the score (each ranging from 0 to 3) of each of a 10-item questionnaire.
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Score on a scale
  Visit 1 (n=114) | 13.55 (7.27)
  Visit 2 (n=99) | 8.75 (6.4)
  Visit 3 (n=91) | 5.46 (5.55)
  Visit 4 (n=79) | 4.89 (6.07)
  Visit 5 (n=76) | 4.18 (6.11)
  Visit 6 (n=69) | 5.39 (6.81)

11. Secondary Outcome: Number of Participants With Satisfactory Health Status
Description: Participant's opinion on his/her health status, as assessed by the following question: "Think about all the ways your psoriasis is affecting you, do you consider that your current status is satisfactory? (Yes/No)"
Time Frame: Week 0 (Visit 1), Week 2 (Visit 2), Week 6 (Visit 3), Week 14 (Visit 4), Week 22 (Visit 5), Week 30 (Visit 6)
Population: Per protocol analysis.
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 124
Participants
  Visit 1 (n=118) | 9
  Visit 2 (n=98) | 42
  Visit 3 (n=94) | 61
  Visit 4 (n=83) | 61
  Visit 5 (n=77) | 63
  Visit 6 (n=68) | 46

ADVERSE EVENTS:
Description: All 133 participants enrolled in the study were included in the safety population.
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 17/133
Other Adverse Events (participants affected / at risk) | 0/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=133)
Coronary artery disease (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Oral pruritus (Gastrointestinal disorders) | 1 (1)
Palatal oedema (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1)
Tuberculosis test positive (Investigations) | 1 (1)
Weight decreased (Investigations) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Syncope vasovagal (Nervous system disorders) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to publication or presentation (abstract, poster, oral communication and any other support existing or future), a copy of the final text should be forwarded by the Investigator(s) to the sponsor, for comment and authorization. Such comments and authorization shall aim to ensure the scientific content of the proposed publication and/or presentations and shall ensure that data and the material referring to the sponsor activities receive fair, accurate, and reasonable presentation.